CLINICAL TRIAL: NCT07401121
Title: Koanewa: A First in Human, Phase 1b, Open-label, Non-randomised, Single Dose Study to Assess the Safety and Tolerability of CTx1000 in Participants Diagnosed With Amyotrophic Lateral Sclerosis
Brief Title: Safety and Tolerability Study of CTx1000 In Participants With Amyotrophic Lateral Sclerosis
Acronym: KOANEWA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celosia Therapeutics Pty Ltd (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALS-AAV9
Record Dates: First submitted 2025-12-10; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
Keywords: CTx1000; gene therapy; motor neuron disease; genetic medicine; Lou Gehrig disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active drug-CTx1000 (Experimental): All participants will receive only one dose of the study drug
  Interventions: Drug: AAV9 Gene therapy

INTERVENTIONS:
Drug: AAV9 Gene therapy — Single dose gene therapy

SUMMARY:
This clinical study is in participants with Amyotrophic Lateral Sclerosis and is designed to evaluate the safety and tolerability of the gene therapy CTx1000.

DETAILED DESCRIPTION:
CTx1000 is an investigational gene therapy that encodes a degron for targeted degradation of TDP-43 following a single dose intra cisterna magna (ICM) delivery in participants diagnosed with Amyotrophic Lateral Sclerosis (ALS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS in accordance with the revised El Escorial criteria and TRICALS risk score
* An overall disease duration of ≤ 2 years after the participant's first symptoms
* No or low circulating anti-AAV9 antibodies (titre ≤ 1:50
* Stable dosing with a standard of care ALS medication (eg, riluzole and edaravone) and other prescription medications for 30 days prior to Screening
* Not pregnant or breastfeeding, or willing to cease breastfeeding
* All participants must use a barrier method of contraception

Exclusion Criteria:

* Any participants with genetic forms of ALS, including C9ORF72 repeat carriers, except for TARDBP gene variants, as confirmed by previous clinical history genetic testing
* Any history of myocardial infarction or stroke within 6 months prior to Screening, or uncontrolled diabetes (HbA1C > 9%)
* Positive test for cytomegalovirus, hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), human immunodeficiency virus (HIV) antibody.
* Inadequate organ function
* Any participant with a current open tracheostomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of CTx1000 in ALS diagnosed participants | 52 weeks
  Incidence of Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interests (AESIs)

SECONDARY OUTCOMES:
To evaluate the long-term safety and tolerability of CTx1000 in ALS diagnosed participants | 3 years
  Incidence of Treatment Emergent Adverse Events (TEAEs), Severe Adverse Events (SAEs) and Adverse Events of Special Interests (AESIs)
To evaluate the long-term pharmacodynamics and immunogenicity of CTx1000 in ALS diagnosed participants | 3 years
  Changes in pre-dose biomarkers (Neurofilament light) in cerebrospinal fluid and anti-drug antibody (ADA)
To evaluate the long-term efficacy of CTx1000 in ALS diagnosed participants | 3 years
  Changes (reduction) from pre-dose Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R)

CONTACTS AND LOCATIONS:
Locations (1):
- Macquarie University Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://celosiatx.com/